CLINICAL TRIAL: NCT05517356
Title: PRospective Study of tailOred Management Strategies fOr Acute Type A Aortic Dissection complicatEd With Malperfusion Syndrome (PROMOTE)
Brief Title: Prospective Study of Tailored Management Strategies for Malperfusion Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Xijie Wu, Director, Head of Cardiosurgery, Clinical Professor, Xiamen Cardiovascular Hospital, Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022YLK19
Record Dates: First submitted 2022-08-16; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Aortic Dissection
Keywords: Tailored management strategies; Aortic dissection; Malperfusion syndrome; Central repair; Endovascular reperfusion.
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malperfusion Cohort (Experimental): Patients presenting to hospital with ATAAD meeting criteria for malperfusion syndrome which includes both components:
  1. Radiographic findings reveal occlusion of the corresponding arteries (including either coronary artery, either carotid artery, celiac trunk, superior mesenteric artery or either iliac artery).
  2. Clinical features of end organ ischemia (abnormal left ventricular wall motion, disorder of consciousness or paralysis, abdominal pain, distended abdomen, pulselessness, loss of sensory or motor function of the lower extremities) OR Laboratory findings suggestive of end organ ischemia (elevated troponin, elevated creatine kinase, lactic acidosis, elevated myoglobin).
  Interventions: Procedure: Tailored management strategies

INTERVENTIONS:
Procedure: Tailored management strategies — Our basic surgical strategies for the central repair operations for ATAAD are as follows. As arterial lines for cardiopulmonary bypass, side branches of the axillary and femoral arteries were used. Circulatory arrest was established when the nasopharyngeal temperature reached 25°C. Anterograde selective cerebral perfusion was performed through the right axillary artery, and the brain was perfused at approximately 5 mL/kg/min. The extent of aortic replacement was determined according to the extent of dissection involvement.
  For malperfused patients with symptom onset within 6 hours, the immediate central repair was performed followed by repeat CTA postoperatively, and endovascular reperfusion was applied if the malperfusion persisted. While for patients with symptom onset beyond 6 hours, delayed central repair were performed after the organ functions improved.

SUMMARY:
Management strategy of malperfusion syndrome in acute type A aortic dissection (ATAAD) patients remains controversial, with different views on when the surgery should be offered. At present, the mortality of ATAAD patients complicated with malperfusion is stubbornly high.

The purpose of this study is to improve the outcomes of ATAAD with malperfusion syndrome. The investigators formulated tailored management strategies for malperfused patients based on the duration of symptoms onset.

DETAILED DESCRIPTION:
ATAAD complicated with malperfusion syndrome Malperfusion syndrome is the most devastating complication of acute type A aortic dissection (ATAAD), which has a poor clinical outcome and has operative mortality ranging from 29% to 89%. However, different views on management of malperfusion exist, with debating on addressing the dissection or the organ malperfusion in priority.

Current different treatment strategies for ATAAD with malperfusion syndrome Immediate central repair, restoration of true lumen flow and depressurization of the false lumen, is the most widely practiced approaches for treating ATAAD regardless of malperfusion syndrome. Nevertheless, with very high operative mortality by the conventional approach for patients with malperfusion, several studies have suggested that patients undergo endovascular reperfusion first until the malperfusion resolves, followed by delayed central repair. This strategy has produced better outcomes for patients, however, it also carries risks of interim mortality due to aortic rupture or multiple-organ failure before central repair. Moreover, a recent study suggested an alternative strategy, which performed aortic surgery and endovascular reperfusion in a hybrid approach for static malperfusion or dynamic malperfusion symptoms more than 6 hours symptoms onset. This alternative strategy improved outcomes with a mortality rate of 16.7%, which was still a little bit high. Overall, the outcomes of ATAAD patients with malperfusion syndrome still need to be improved.

Tailored management strategies The tailored management strategies were: for malperfused patients with symptom onset within 6 hours, the immediate central repair was performed followed by repeat CTA postoperatively, and endovascular reperfusion was applied if the malperfusion persisted. While for patients with symptom onset beyond 6 hours, delayed central repair were performed after the organ functions improved.

Study Rationale As noted above, malperfusion syndrome is a rapidly lethal condition that every cardiovascular surgeon is faced with at some point. Despite the optimization of approaches for ATAAD presented with malperfusion in recent years, there appears to be some room to improve our outcomes even further. The investigators believe that the tailored management strategies, which aimed at reducing the duration of end-organ ischemia, may provide a promising treatment option for these patients. However, further prospective study and follow-up data are necessary to confirm the efficacy and safety of this new strategy.

ELIGIBILITY:
Inclusion Criteria:

* Acute type A aortic dissection is confirmed by CTA;
* The symptoms onset time < 2 weeks;
* Patients diagnosed with an ATAAD , with a new diagnosis of malperfusion syndrome, by meeting both of the following criteria:

  1. Radiographic findings reveal occlusion of the corresponding arteries (including either coronary artery, either carotid artery, celiac trunk, superior mesenteric artery or either iliac artery)
  2. Clinical features of end organ ischemia (abnormal left ventricular wall motion, disorder of consciousness or paralysis, abdominal pain, distended abdomen, pulselessness, loss of sensory or motor function of the lower extremities) OR Laboratory findings suggestive of end organ ischemia (elevated troponin, elevated creatine kinase, lactic acidosis, elevated myoglobin).

Exclusion Criteria:

* The branch arteries did not involved by ATAAD (non-malperfusion);
* Patients presented with bloody stools or melena on admission;
* Patients presented with bilaterally fixed dilated pupils, hemorrhagic infarction or herniation of brain;
* Patients and (or) their families refused surgery;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality (number of all cause death) | 12 months
  All cause death

SECONDARY OUTCOMES:
Low cardiac output syndrome | 30 days
  Number of participants complicated with low cardiac output syndrome after surgery
New cerebrovascular events | 30 days
  Number of participants complicated with new cerebrovascular events after surgery
Intestinal necrosis | 30 days
  Number of participants complicated with intestinal necrosis after surgery
Lower limb necrosis | 30 days
  Number of participants complicated with lower limb necrosis after surgery
Multiple organ failure | 30 days
  Number of participants complicated with multiple organ failure after surgery
Extracorporeal membrane oxygenation | 30 days
  Number of participants requiring extracorporeal membrane oxygenation after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiac Surgery, Xiamen Cardiovascular Hospital of Xiamen University, School of Medicine, Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deeb GM, Williams DM, Bolling SF, Quint LE, Monaghan H, Sievers J, Karavite D, Shea M. Surgical delay for acute type A dissection with malperfusion. Ann Thorac Surg. 1997 Dec;64(6):1669-75; discussion 1675-7. doi: 10.1016/s0003-4975(97)01100-4. PMID 9436553
- [Background] Geirsson A, Szeto WY, Pochettino A, McGarvey ML, Keane MG, Woo YJ, Augoustides JG, Bavaria JE. Significance of malperfusion syndromes prior to contemporary surgical repair for acute type A dissection: outcomes and need for additional revascularizations. Eur J Cardiothorac Surg. 2007 Aug;32(2):255-62. doi: 10.1016/j.ejcts.2007.04.012. Epub 2007 May 17. PMID 17500002
- [Background] Girdauskas E, Kuntze T, Borger MA, Falk V, Mohr FW. Surgical risk of preoperative malperfusion in acute type A aortic dissection. J Thorac Cardiovasc Surg. 2009 Dec;138(6):1363-9. doi: 10.1016/j.jtcvs.2009.04.059. Epub 2009 Sep 5. PMID 19733865
- [Background] Ahmed Y, van Bakel PAJ, Patel HJ. Addressing malperfusion first before repairing type A dissection. JTCVS Tech. 2021 May 4;10:1-5. doi: 10.1016/j.xjtc.2021.04.029. eCollection 2021 Dec. No abstract available. PMID 34977693
- [Background] Fann JI, Sarris GE, Mitchell RS, Shumway NE, Stinson EB, Oyer PE, Miller DC. Treatment of patients with aortic dissection presenting with peripheral vascular complications. Ann Surg. 1990 Dec;212(6):705-13. doi: 10.1097/00000658-199012000-00009. PMID 2256762
- [Background] Ehrlich MP, Ergin MA, McCullough JN, Lansman SL, Galla JD, Bodian CA, Apaydin A, Griepp RB. Results of immediate surgical treatment of all acute type A dissections. Circulation. 2000 Nov 7;102(19 Suppl 3):III248-52. doi: 10.1161/01.cir.102.suppl_3.iii-248. PMID 11082396
- [Background] Girardi LN, Krieger KH, Lee LY, Mack CA, Tortolani AJ, Isom OW. Management strategies for type A dissection complicated by peripheral vascular malperfusion. Ann Thorac Surg. 2004 Apr;77(4):1309-14; discussion 1314. doi: 10.1016/j.athoracsur.2003.09.056. PMID 15063257
- [Background] Uchida K, Karube N, Kasama K, Minami T, Yasuda S, Goda M, Suzuki S, Imoto K, Masuda M. Early reperfusion strategy improves the outcomes of surgery for type A acute aortic dissection with malperfusion. J Thorac Cardiovasc Surg. 2018 Aug;156(2):483-489. doi: 10.1016/j.jtcvs.2018.02.007. Epub 2018 Feb 13. PMID 29548594
- [Background] Yang B, Rosati CM, Norton EL, Kim KM, Khaja MS, Dasika N, Wu X, Hornsby WE, Patel HJ, Deeb GM, Williams DM. Endovascular Fenestration/Stenting First Followed by Delayed Open Aortic Repair for Acute Type A Aortic Dissection With Malperfusion Syndrome. Circulation. 2018 Nov 6;138(19):2091-2103. doi: 10.1161/CIRCULATIONAHA.118.036328. PMID 30474418
- [Background] Chiu P, Tsou S, Goldstone AB, Louie M, Woo YJ, Fischbein MP. Immediate operation for acute type A aortic dissection complicated by visceral or peripheral malperfusion. J Thorac Cardiovasc Surg. 2018 Jul;156(1):18-24.e3. doi: 10.1016/j.jtcvs.2018.01.096. Epub 2018 Feb 21. PMID 29615333
- [Background] Tsagakis K, Janosi RA, Frey UH, Schlosser T, Chiesa R, Rassaf T, Jakob H. True Lumen Stabilization to Overcome Malperfusion in Acute Type I Aortic Dissection. Semin Thorac Cardiovasc Surg. 2019 Winter;31(4):740-748. doi: 10.1053/j.semtcvs.2018.11.012. Epub 2018 Dec 8. PMID 30529161